CLINICAL TRIAL: NCT07174232
Title: Cross-training of Russian Current and Muscle Energy Techniques on Pain, Muscle Strength, and Functional Disabilities in Circumferential Upper Arm Burn
Brief Title: Russian Current and Muscle Energy Techniques on Circumferential Upper Arm Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005677
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: RCT,prospective
Who Masked: Participant
Masking Description: single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Russian current and muscle energy techniques (Experimental): Muscle energy technique Plus Russian Current
  Interventions: Other: Russian current and muscle energy techniques
- Russian Current (Experimental): Russian Current application
  Interventions: Other: Russian Current
- Control (No Intervention): No intrtvention

INTERVENTIONS:
Other: Russian current and muscle energy techniques — The participants will have the electrodes placed on their biceps and triceps muscles for the Russian current treatment and were positioned comfortably, typically in a supine or seated position, depending on the muscle group being targeted. This positioning ensured stability and allowed for the effective application of the MET .
  Arms: Russian current and muscle energy techniques
Other: Russian Current — The participants will have the electrodes placed on their biceps and triceps muscles for the Russian current treatment. For the biceps, one electrode will be placed on the middle of the muscle, about halfway between the shoulder and elbow, while the second electrode will be placed slightly above it, closer to the shoulder
  Arms: Russian Current

SUMMARY:
Burn injuries, particularly circumferential upper arm burns, present significant challenges in rehabilitation due to their impact on pain management, muscle strength, and overall functional abilities. These injuries can lead to severe scarring and contractures, which further complicate the recovery process and affect the patient's quality of life. Traditional rehabilitation approaches often fall short in addressing the multifaceted needs of burn survivors, necessitating the exploration of innovative therapeutic techniques.

DETAILED DESCRIPTION:
Russian current, a form of electrical stimulation, has been extensively utilized in physical therapy to enhance muscle strength and reduce muscle atrophy. Its application in burn rehabilitation is promising due to its ability to stimulate muscle contractions, thereby aiding in maintaining muscle mass and strength. When applied to patients with circumferential upper arm burns, Russian current can potentially mitigate the decline in muscle function while alleviating pain. This method not only supports the physical recovery process but also contributes to improved overall patient well-being by reducing discomfort and enhancing functional capabilities.

Muscle energy techniques (MET), on the other hand, are manual therapy interventions designed to improve muscular flexibility and range of motion. By engaging the patient's own muscle contractions against a counterforce, MET can effectively reduce muscle tightness and improve joint function. When integrated with Russian current, MET can offer a comprehensive rehabilitation strategy for patients with upper arm burns. This cross-training approach aims to synergistically improve outcomes by addressing pain management, muscle strength recovery, and functional disability reduction, ultimately leading to a more holistic recovery process for burn survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years,
* Unilateral circumferential elbow and upper arm burn requiring rehabilitation,
* Medical stability for physical therapy interventions,
* The ability to provide informed consent

Exclusion Criteria:

* Neurological disorders, severe cognitive impairment, contraindications to electrical stimulation,
* Recent upper limb surgery
* Pregnant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Muscle power test | at baseline and at 12 weeks
  Using a Biodex System 3 PRO dynamometer (Biodex Medical Systems, Shirley, New York).Measurements will be taken before and after the 12-week treatment period. The peak torque (PT) of the biceps and triceps muscles was measured in Newton meters (Nm) for the dominant (affected) side

SECONDARY OUTCOMES:
Visual Analogue Scale | at baseline and at 12 weeks
  A visual analogue scale (VAS) is a measurement instrument used in health and medicine to quantify subjective experiences like pain or fatigue on a simple line, with 1 end representing the least intense sensation and 10 the most intense.
Upper-Extremity Disability: (DASH) questionnaire | at baseline and at 12 weeks
  The DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire is a 30-item, self-report tool used to measure physical function and symptoms in people with upper-limb musculoskeletal disorders.The questionnaire score ranges from 0 to 100, where 0 indicates no disability and 100 represent the most severe disability

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt